



# BPIT Clinical Study: Statistical Analysis Plan Summary (Version 1.1)

**Focus:** Interpreting Patient Outcomes and Clinical Efficacy **Date:** November 25, 2025 | **Protocol:** BPIT Multi-Site Clinical Study v3.2 **Principal Investigator:** Dr. Neeraj Mehta, PhD | **Study ID:** MACREB-BPIT-2025-014 **Anticipated Analysis Date:** Post-Data Lock (February 2026)

## **Version History:**

- Version 1.0: Initial plan, November 6, 2025.
- Version 1.1: Reviewed for ClinicalTrials.gov submission on November 25, 2025; no changes to analysis methods or criteria.

## 1. Study Goals and Outcome Measures

This analysis plan is designed to rigorously determine if the **BPIT intervention** delivers clinically meaningful benefits in movement, pain, and function compared to a standard progressive overload protocol.

| Measure Category | Key Clinical Measure | Goal/Success Criteria (Hypothesis) | Clinical Relevance |
|---|---|---|---|
| Primary Efficacy | Movement Efficiency<br>Score (MES, 0–10):<br>Change from baseline<br>(Week 0) to<br>end-of-study (Week 5). | BPIT must improve MES by \ge 25% (Statistically significant, p<0.05). | A simple, validated metric for overall biomechanical function and movement quality. The primary indicator of treatment success. |
| Secondary Outcomes | Range of Motion<br>(ROM) (degrees) | Improvement of 15–20%. | Direct measure of joint/tissue flexibility and mobility. |
| | VAS Pain Score<br>(0–10) | Reduction of \approx <b>40%</b> . | Pain relief is a critical patient-reported outcome. |
| | Strength Index (Reps<br>\times Load) | Increase of 20–30%. | Objective measure of functional capacity and muscular performance. |
| | Mobility Limitation<br>(%) | Reduction of \approx <b>25%</b> . | How the change in<br>MES/ROM translates to |





| Measure Category | Key Clinical Measure | Goal/Success Criteria | Clinical Relevance |
|---|---|---|---|
| | | (Hypothesis) | |
| | | | daily functional tasks. |
| Exploratory | Heart Rate Variability | Increase of \approx | A biomarker for |
| | (HRV - RMSSD) | 10%. | autonomic nervous |
| | | | system health and |
| | | | recovery. |

#### 2. La Enrollment & Statistical Power

The study is adequately powered to detect clinically relevant changes.

- **Target Enrollment:** \mathbf{n=116} total participants (58 in BPIT group, 58 in Control group).
- **Completers:** Aiming for 100 participants after accounting for \approx 10–14% expected dropout.
- Statistical Assurance: We have an 80% chance (Power) of detecting a moderate but clinically important difference (Cohen's d=0.5).
- **Minimum Detectable Change:** The study is structured to confirm if BPIT delivers at least an **18% change in MES**. If the improvement is less than this, we will likely not be able to declare it statistically superior.

## 3. III Interpretation of Key Analyses

We will use standard statistical methods appropriate for pre-post and group comparisons.

| Clinical Question | Statistical Approach | Measures Involved | Clinical Interpretation of |
|---|---|---|---|
| | | | Results |
| Did the BPIT | Paired t-test (or | Wk 0 vs. Wk 5 MES | If p<0.05, the treatment |
| treatment work? | Non-Parametric | change (within the | caused a significant |
| | alternative). | BPIT group). | improvement in |
| | | | movement efficiency for |
| | | | the participants. |
| Is BPIT better than | Independent | BPIT vs. Control | If p<0.05, the BPIT |
| standard care? | t-test/ANOVA | (comparing the change | protocol is superior to |
| | (Between-Group). | scores). | the control intervention |
| | | | in improving the |
| | | | outcomes. |
| How did patients | Repeated-Measures | ROM, VAS, Strength | Helps determine the |
| progress over time? | ANOVA. | across Wk 0, Wk 3, and | speed and |
| | | Wk 5. | maintenance of clinical |
| | | | effect. Post-hoc |





| Clinical Question | Statistical Approach | Measures Involved | Clinical Interpretation of |
|---|---|---|---|
| | | | Results |
| | | | analysis (e.g., Tukey) |
| | | | will pinpoint when the |
| | | | significant changes |
| | | | occurred. |
| What predicts the | Multiple Linear | BPIT Line (1-5 score), | Identifies clinical |
| best response? | Regression. | Age, Gender predicting | predictors—e.g., if a |
| | | MES change. | high score on the "BPIT |
| | | | Line 3" movement |
| | | | pattern is most |
| | | | associated with |
| | | | success. |
| Is the treatment safe? | Chi-Square/Fisher's | Adverse Event (AE) | Confirms there is <b>no</b> |
| | Exact Test. | frequency by | difference in safety |
| | | group/site. | risk (AEs) between the |
| | | | BPIT and control |
| | | | protocols. |

**IMPORTANT NOTE:** Due to testing multiple secondary outcomes, we will use a **Bonferroni Adjustment** (p<0.0125 required for secondary outcomes) to maintain the integrity of the results. Clinicians should focus on the **Effect Size** (**Cohen's d**) and the **95% Confidence Interval** (**CI**) in addition to the p-value, as these indicate the *magnitude* and *precision* of the clinical benefit.

## 4. Data Quality and Reporting

- **Missing Data Plan:** If a participant misses an assessment (e.g., Week 5), we will use their **Last Observation Carried Forward (LOCF)** for the final analysis, *unless* more than 10% of the data is missing, in which case we will conduct a separate sensitivity analysis.
- Final Outputs: Results will be summarized in clinically relevant tables (e.g., Means \pm SD) and figures (e.g., Box Plots showing MES improvement and Spider Charts for the five BPIT "Lines").

Date: November 25, 2025

Reviewed and Approved by:

Dr. Neeraj Mehta, PhD Dr Santa March, PhD Dr Anupama Mahagan, PhD MACREB Statistics Consultant